CLINICAL TRIAL: NCT00704522
Title: Evaluation of Adherence Rate in Patients Receiving PegIntron Pen / Rebetol for Hepatitis C in Conjunction With a Patient Assistance Program.
Brief Title: Adherence in Patients Receiving PegIntron Pen/Rebetol for Hepatitis C in Conjunction With a Patient Assistance Program (Study P04281)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04281
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with hepatitis C: Patients receiving a patient assistance program during therapy for hepatitis C at sites in Austria.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908); Behavioral: Patient assistance program

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: PegIntron, PegIntron pen
Drug: Ribavirin (SCH 18908) — Peginterferon alfa-2b and ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol
Behavioral: Patient assistance program — Assistance programs will be classified as follows:
  1. Medications used prophylactically or for treatment(Growth factors: RBC and neutrophil; Psychiatric medications; Other medications)
  2. Other interventions (Psychotherapy, Patient Support Groups, Visiting Nurse, Nurse Telephone Calls, Nurse support in office, Other health care professional support, Educational Literature).
  In Austria, sites with adherence nurses and side effect handouts will be compared with sites using side effect handouts only.

SUMMARY:
Patients receiving a patient assistance program during therapy for Hepatitis C will be enrolled into this study. All patients will receive PegIntron pen and Rebetol according to label and the patient assistance program. This study will be compared to similar studies from other clinics using various patient support programs for the purpose of designing future comparative phase IV studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hepatitis C

Exclusion Criteria:

* According to the products' labeling (refer to Warnings, contraindications, and safety sections).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving a patient assistance program during therapy for hepatitis C at sites in Austria.
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- PegIntron Pen/Rebetol Without Patient Assistance Program: PegIntron & Rebetol will be administered according to the products' labeling.
- PegIntron Pen/Rebetol With Patient Assistance Program: PegIntron & Rebetol will be administered according to the products' labeling. Assistance programs include medications used prophylactically or for treatment (Growth factors: RBC and neutrophil; Psychiatric medications; Other
  medications) - Other interventions (Psychotherapy, Patient Support Groups, Visiting Nurse, Nurse Telephone Calls, Nurse support in office, Other health care professional support, Educational Literature).
Period: Overall Study
Arm/Group | PegIntron Pen/Rebetol Without Patient Assistance Program | PegIntron Pen/Rebetol With Patient Assistance Program
Started | 481 | 120
Completed | 298 | 75
Not Completed | 183 | 45
Not completed — Lack of Efficacy | 65 | 17
Not completed — Failure to appear again at hospital | 56 | 10
Not completed — Withdrawal by Subject | 17 | 8
Not completed — Adverse Event | 9 | 1
Not completed — Undefined causes | 9 | 7
Not completed — No information on therapy end | 27 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIntron Pen/Rebetol Without Patient Assistance Program | PegIntron Pen/Rebetol With Patient Assistance Program | Total
Number analyzed (Participants) | 481 | 120 | 601
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.85 (12.98) | 41.38 (11.96) | 41.76 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 42 | 217
  Male | 306 | 78 | 384
Region of Enrollment [Number; unit: participants]
  Austria | 481 | 120 | 601

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Treatment With PegIntron Pen/Rebetol Therapy for Hepatitis C When Administered With a Patient Assistance Program
Time Frame: 24 or 48 weeks (depending on genotype) and 24 weeks of follow up
Population: All participants
Measure: Number; unit: Participants
Arm/Group | PegIntron Pen/Rebetol Without Patient Assistance Program | PegIntron Pen/Rebetol With Patient Assistance Program
Number analyzed (Participants) | 481 | 120
Participants | 298 | 75

2. Primary Outcome: Average Length of Treatment With PegIntron/Rebetol
Time Frame: After start of treatment
Population: Number of participants who received study drug
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | PegIntron Pen/Rebetol Without Patient Assistance Program | PegIntron Pen/Rebetol With Patient Assistance Program
Number analyzed (Participants) | 478 | 119
Weeks | 28.8 (14.6) | 27.3 (14.7)

ADVERSE EVENTS:
Description: Population for Adverse Event reporting is based on all participants who received study drug (N=597).
Arm/Group | PegIntron Pen/Rebetol
Serious Adverse Events (participants affected / at risk) | 20/597
Other Adverse Events (participants affected / at risk) | 100/597
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Pen/Rebetol (N=597)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
INJECTION SITE REACTION (General disorders) | 1 (1)
ABSCESS SWEAT GLAND (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
TUBERCULOSIS (Infections and infestations) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1)
SMEAR CERVIX ABNORMAL (Investigations) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MYELOPATHY (Nervous system disorders) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron Pen/Rebetol (N=597)
ANAEMIA (Blood and lymphatic system disorders) | 49 (50)
LEUKOPENIA (Blood and lymphatic system disorders) | 43 (51)
DEPRESSION (Psychiatric disorders) | 38 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No